CLINICAL TRIAL: NCT04316286
Title: Telemedicine With Mobile Internet Devices for Innovative Multidisciplinary Patient-centred Care of Patients With Narcolepsy
Brief Title: TElemedicine for NARcolepsy
Acronym: TENAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Usl di Bologna (Other Government)
Collaborators: University of Bologna (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); IRCCS Istituto delle Scienze Neurologiche di Bologna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RF-2016-02364742
Record Dates: First submitted 2020-01-30; First posted 2020-03-20 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Narcolepsy
MeSH Terms: conditions — Narcolepsy | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-multidisciplinary participants (Experimental): Patients undergoing televisit
  Interventions: Procedure: Tele-multidisciplinary care
- In-office standard participants (Other): Patients undergoing in-office visits
  Interventions: Other: Standard care

INTERVENTIONS:
Procedure: Tele-multidisciplinary care — Scheduled televisit by sleep medicine specialists, endocrinologists, legal-medicine specialists
  Arms: Tele-multidisciplinary participants
Other: Standard care — Scheduled in-office visit by sleep medicine specialists, endocrinologists, legal-medicine specialists
  Arms: In-office standard participants

SUMMARY:
The TENAR trial is the first randomized controlled trial (RCT) designed to evaluate the feasibility, efficacy, safety, and costs of a Telemedicine multidisciplinary approach for the management of narcolepsy.

Open RCT assessing the non-inferiority of the multidisciplinary management of narcolepsy via Video Consultation (VC) through Mobile Telemedicine devices compared to usual in-office care. 202 children and adults with narcolepsy will be randomly allocated in 1:1 ratio to VC or in-office usual care for a 12 months follow-up. At baseline, all patients will undergo a neurologic, metabolic, and psychosocial assessment. Primary (i.e., excessive daytime sleepiness according to the Epworth Sleepiness Scale) and secondary endpoints (i.e., other symptoms, metabolic control, quality of life, patient and family satisfaction with care, feasibility, safety, and costs) will be measured at 6 and 12 months. The investigators expect the Telemedicine approach not only to be non-inferior for sleepiness control but also to significantly improve other patient-centred outcomes compared to the usual in-office care.

ELIGIBILITY:
Inclusion Criteria:

• Adolescents (≥14 years old) and adults with a diagnosis of narcolepsy according to ICSD-3 criteria at their first ("incident") or with established diagnosis ("prevalent" subjects), able to provide consent

Exclusion Criteria:

* inability to read, write, or using a tablet;
* major psychiatric disorders.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-11-24 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
excessive daytime sleepiness | 12 months
  Measured by the Epworth Sleepiness Scale. The Epworth Sleepiness Scale is a self-administered form with eight items investigating sleep propensity in different real-life situations during the preceding months. Each item can received 0-3 points, thus the final score ranges from 0 (best score) to 24 (worse score). The proposed range for normal subjects is 0-10

SECONDARY OUTCOMES:
metabolic control - weight Changes | 12 months
  metabolic control - weight Changes of weight in kilograms. [Time frame: 12 months]
metabolic control - lipid profile Changes | 12 months
  metabolic control - lipid profile Changes of: total cholesterol; high-density lipoprotein cholesterol; low-density lipoprotein cholesterol; total triglycerides. All are measured in milligrams per deciliter (mg/dl).
  [Time frame: 12 months]
metabolic control - glycemic profile Changes | 12 months
  metabolic control - glycemic profile Changes of fasting glycemia measured in milligrams per deciliter (mg/dl). [Time frame: 12 months]
metabolic control - caloric intake Changes | 12 months
  metabolic control - caloric intake Changes of caloric intake measured by a food diary. [Time frame: 12 months]
metabolic control - physical activity Changes | 12 months
  metabolic control - physical activity Changes of physical activity measured by the International Physical Activity Questionnaire (IPAQ). Total physical activity is measured in MET-min/week and time spent sitting, and it is ranked in three levels: low; moderate; high.
  [Time frame: 12 months]
quality of life - Short-Form 36-Item Questionnaire | 12 months
  Quality of life - Short-Form 36-Item Questionnaire (SF-36) Changes of SF-36 health related quality of life (HRQOL) scales. This tool presents 36 questions. Eight health domains are assessed (physical activities; social activities; limitations in role activities because of physical health problems; bodily pain; mental health; limitations in role activities because of emotional problems; vitality; general health perceptions). Each domain measures a level of HRQOL with a scale between 0-100, with 0 being bad quality of life and 100 being good.
  [Time frame: 12 months]
quality of life - Pediatric Quality of Life Inventory | 12 months
  Quality of life - Pediatric Quality of Life Inventory (PedsQL) Changes of PedsQL health related quality of life (HRQOL) scales. This is a tool of 23 questions comprising four generic domains: physical functioning; emotional functioning; social functioning; school functioning. These domains are measured by a 0-100 scale. Higher scores indicate better HRQOL.
  [Time frame: 12 months]
patient and family satisfaction with care | 12 months
  patient and family satisfaction with care, measured by an ad-hoc devised form (named Co-Tenar), assessing qualitatively the satisfaction level.
safety | 12 months
  safety, in terms of number (percent) of full drop-outs, partial drop-outs (patients changing procedure), adverse reactions to drugs in both group of intervention (standard in-office visit arm, video-consultation arm).
costs | 12 months
  costs related to the disease management (drugs, tests, hospitalization, journeys) will be assessed, by means of a standardized interview, in both group of intervention (standard in-office visit arm, video-consultation arm).

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Plazzi, Principal Investigator — IRCCS Istituto delle Scienze Neurologiche di Bologna
Locations (1):
- Irccs - Istituto Delle Scienze Neurologiche, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ingravallo F, Vignatelli L, Pagotto U, Vandi S, Moresco M, Mangiaruga A, Oriolo C, Zenesini C, Pizza F, Plazzi G. Protocols of a diagnostic study and a randomized controlled non-inferiority trial comparing televisits vs standard in-person outpatient visits for narcolepsy diagnosis and care: TElemedicine for NARcolepsy (TENAR). BMC Neurol. 2020 May 11;20(1):176. doi: 10.1186/s12883-020-01762-9. PMID 32393279